CLINICAL TRIAL: NCT00453739
Title: TVT-World Wide Observational Registry for Long-Term Data
Brief Title: TVT Worldwide Registry
Status: Completed | Type: Observational
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 300-06-006
Record Dates: First submitted 2007-03-28; First posted 2007-03-29 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-05

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The objective of this observational study is to obtain long -term clinical and patient reported outcomes on the use of the GYNECARE family of TVT (Tension-Free Vaginal Tape) systems in women with stress urinary incontinence.

DETAILED DESCRIPTION:
Sites may include patients with either the GYNECARE TVT SECUR System, GYNECARE TVT System, or the GYNECARE TVT Obturator System

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with SUI who are suitable candidates for a TVT system, as according the relevant Instructions for Use (IFU).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with SUI who are suitable candidates for a TVT system, according the relevant Instructions for Use (IFU).
Sampling Method: Non-Probability Sample
Enrollment: 1407 (Actual)
Dates: Start 2007-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Standing cough stress test | 12 months

SECONDARY OUTCOMES:
I-QOL score | 3, 6, 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: David Robinson, MD, Study Director — Ethicon, Inc.
Locations (30):
- United States (15):
  - Southern California Permanente Medical Group, Downey, California
  - Milestone Medical Research, Englewood, Colorado
  - Specialists in Urology, Naples, Florida
  - Illinois Urogynecology LTD, Oak Lawn, Illinois
  - Michigan Institute of Women's Health, Dearborn, Michigan
  - Women's Health Center of West Michigan, Grand Rapids, Michigan
  - Female Pelvic Medicine & Reconstructive Surgery, Minneapolis, Minnesota
  - Sheldon J. Freedman MD, Las Vegas, Nevada
  - University of Rochester OB/Gyn Department, Rochester, New York
  - Seton Center, Good Samaritan Hospital, West Chester, Ohio
  - The Institute for Female Pelvic Medicine and Reconstructive Surgery, Allentown, Pennsylvania
  - Advanced Clinical Concepts, West Reading, Pennsylvania
  - Vanderbilt University Medical School, Nashville, Tennessee
  - Northern Virginia Pelvic Surgery Associates, Annandale, Virginia
  - Sound Urological Associates, Edmonds, Washington
- Australia (3):
  - The Townsville Hospital Department of Urogynaecology, Douglas
  - Gold Coast Health Service, Southport
  - Queen Elizabeth Hospital, Woodville
- Abteilung fuer Gynaekologie, Mödling, Austria
- Wentworth-Limeridge Medical Centre, Hamilton, Ontario, Canada
- Universitatsfrauenklinik, Tübingen, Germany
- Kandang Kerbau Women's and Children's Hospital, Singapore, Singapore
- South Africa (3):
  - Kingsbury House, Cape Town
  - Pretoria Urology Hospital, Hatfield
  - Arwyp Hospital, Kempton
- Samsung Medical Center, Seoul, South Korea
- United Kingdom (4):
  - Ulster Hospital Belfast, Belfast
  - Stoke Mandeville Hospital, Buckinghamshire
  - Glasgow Southern General, Glasgow
  - Leicester General Hospital, Leicester

REFERENCES:
- [Result] Tincello DG, Botha T, Grier D, Jones P, Subramanian D, Urquhart C, Kirkemo A, Khandwala S; TVT Worldwide Registry Investigators. The TVT Worldwide Observational Registry for Long-Term Data: safety and efficacy of suburethral sling insertion approaches for stress urinary incontinence in women. J Urol. 2011 Dec;186(6):2310-5. doi: 10.1016/j.juro.2011.07.078. Epub 2011 Oct 20. PMID 22014817